CLINICAL TRIAL: NCT03591341
Title: Melatonin Degradation Rate in Human Milk
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-17-0035-CTIL
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-07

CONDITIONS: Preterm Infant; Lactation
Keywords: melatonin; breast milk
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nursing women: women who gave birth and are breast feeding their baby- melatonin level in pumped breast milk have been checked
  Interventions: Diagnostic Test: melatonin level in pumped breast milk

INTERVENTIONS:
Diagnostic Test: melatonin level in pumped breast milk — diagnostic test of melatonin level in pumped breast milk

SUMMARY:
Our long term hypothesis is that giving premature infants breast milk that was pumped during the night and has high concentration of melatonin will improve outcome of several clinical conditions related to premature infants. Prior to testing this, we need to learn the pharmacokinetics of melatonin in vitro.

In this preliminary research we would like to check the levels of melatonin in breast milk pumped during the night, and evaluate the rate of degradation of the melatonin to determine the half life of melatonin in pumped breast milk (in vitro).

DETAILED DESCRIPTION:
The study includes 10 nursing women. Each woman will bring a frozen 5 ml sample of breast milk that was pumped at 03:00 AM. The samples will be collected at the NICU department of Carmel Medical Center and will be stored at deep freeze (-20°C). The samples will be numerically coded and will be kept anonimously. After defrosting the samples, melatonin concentration will be checked in the hospital laboratory every hour, for 4 hours. If meltonin levels will be detectable after 4 hours, continous measurements will be done at 8 hours and at 12 hours after defrosting. The samples will be tested with IBL Melatonin ELISA kit. For control we will use breast milk that was pumped at 10:00 am (when melatonin excretion is minimal). At the end of the analysis the samples will be thrown away.

ELIGIBILITY:
Inclusion Criteria:

1. Women that are breast feeding and will pump and freeze a milk sample at 03:00 AM
2. Women at least one week after delivery

Exclusion Criteria:

1. A sample that will not be freezed right after the pump
2. Women that are taking hypnotic drugs
3. Women that are taking melatonin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only women that gave birth and are breast feeding their babies
Study Population: healthy women who are breast feeding
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
melatonin stability in human milk | 24 hours
  melatonin levels in human milk samples are checked every hour after defrost

CONTACTS AND LOCATIONS:
Overall Officials: michal molad, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen Engler A, Hadash A, Shehadeh N, Pillar G. Breastfeeding may improve nocturnal sleep and reduce infantile colic: potential role of breast milk melatonin. Eur J Pediatr. 2012 Apr;171(4):729-32. doi: 10.1007/s00431-011-1659-3. Epub 2011 Dec 29. PMID 22205210
- [Background] Katzer D, Pauli L, Mueller A, Reutter H, Reinsberg J, Fimmers R, Bartmann P, Bagci S. Melatonin Concentrations and Antioxidative Capacity of Human Breast Milk According to Gestational Age and the Time of Day. J Hum Lact. 2016 Nov;32(4):NP105-NP110. doi: 10.1177/0890334415625217. Epub 2016 Jul 10. PMID 27121237